CLINICAL TRIAL: NCT04449835
Title: The Intracept Global Registry
Brief Title: The Intracept Global Registry ( TIGR ) - Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Pilot Study converted to NCT 05660512 prospective single arm cohort study
Sponsor: Relievant Medsystems, Inc. (Industry)
Collaborators: M Squared Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Zack McCormick, Assistant Professor and Director of Clinical Spine Research, University of Utah
Other Study IDs: CIP 0014
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intracept Procedure — radio frequency ablation of the basivertebral nerve for the relief of chronic vertebrogenic low back pain

SUMMARY:
The Intracept Global Registry is a prospective, noninterventional, observational global post market independent data collection of the ongoing effectiveness, safety, and satisfaction outcomes for patients treated with the Intracept Procedure. This registry will be conducted according to Good Clinical Practice (GCP) guidelines, including participant verbal informed consent and Independent Review Board (IRB) / Ethics Committee (EC) approval and oversight.

Registry design, conduct, analysis, and reporting are overseen by the Principal Investigator (PI) and the cross-specialty TIGR Physician Steering Committee.

DETAILED DESCRIPTION:
Participants in the registry will have seven study visits over a period of five years (one prior to procedure and 6 post their procedure). Study visits will be conducted via telephone by a third-party CRO and independent clinical research coordinators. Participants will be verbally consented and then evaluated via telephonic study visits at baseline (prior to procedure) and at 3, 12, 24, 36, 48, and 60 months post their Intracept Procedure.

Primary and secondary objectives are based on patient reported outcomes for functional improvement, pain reduction, and physical and mental health pre and post procedure. The study will also look at utilization of injections and pain interventions/surgery for treatment of low back pain post Intracept.

ELIGIBILITY:
Inclusion Criteria:

All patients scheduled for the Intracept procedure and whose treating physician is referring to the registry

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have the Intracept procedure and whose treating physician is referring to the registry
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Reduction | 3 months post procedure
  Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 3 months.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) improvement | 3, 12, 24, 36, 48 and 60 months post procedure
  Mean improvement in ODI scores from baseline (scale 0 to 100)
Numeric Pain Score | 3, 12, 24, 36, 48 and 60 months post procedure
  Mean reduction in patient reported low back pain from baseline (scale 0 no pain to 10 worst pain imaginable)
Combined Responder Rates (improvement thresholds of ODI ≥ 15 and NPS ≥ 2) | 3, 12, 24, 36, 48 and 60 months post procedure
  Percent of responders meeting both thresholds
PROMIS 29 Change | 3, 12, 24, 36, 48 and 60 months post procedure
  Mean change in PROMIS-29 from baseline
Injections utilization compared to baseline | 3, 12, 24, 36, 48 and 60 months post procedure
  Numbers of injections post procedure compared to baseline
Post ablation pain interventions/surgeries | 3, 12, 24, 36, 48 and 60 months post procedure
  Numbers of pain interventions/surgeries post procedure compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zachary McCormick, MD, FAAPMR, Principal Investigator — Spine and Pain Medicine, University of Utah School of Medicine
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No